CLINICAL TRIAL: NCT00167232
Title: Naltrexone and Psychosocial Treatments for the Treatment of Cocaine Dependence Complicated by Alcohol Dependence
Brief Title: Naltrexone in Two Models of Psychosocial Treatments for Cocaine and Alcohol Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kyle Kampman, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 57300; P60DA005186 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2013-09

CONDITIONS: Cocaine Dependence; Alcoholism
Keywords: naltrexone; cocaine dependence; alcohol dependence; psychosocial treatment
MeSH Terms: conditions — Cocaine-Related Disorders; Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Naltrexone 150mg/day (Active Comparator)
  Interventions: Drug: Naltrexone
- Placebo Sugar Pill (Placebo Comparator)
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
The purpose of this study is to see whether naltrexone is safe and useful in preventing alcohol relapse, as well as in decreasing craving for alcohol in people with a diagnosis of alcohol and cocaine dependence. Naltrexone is approved by the Food and Drug Administration (FDA) for the treatment of alcohol dependence. However, the medication was not approved as yet at the dosage we will use in this study. The dosage we will use for the study (150 mg), is greater than the recommended dosage from the Physician's Desk Reference (50mg). Unlike other medicines (like Antabuse) useful in the treatment of alcohol dependence, naltrexone will not make you sick if you drink alcohol. Rather, people who are taking this medication have reported that it helps decrease the pleasure associated with drinking for them. This study is being conducted because the medication (Naltrexone) has not been well studied in people with both alcohol and cocaine dependence, so it is still investigational.

We believe that if we can reduce alcohol consumption through naltrexone and psychotherapy, this may lead to reduced cocaine use. We are also conducting this study to test two different types of psychotherapy as a method for reducing cocaine and alcohol use. One type of psychotherapy is designed to help people learn to cope with situations that put them at high risk for relapse to cocaine and/or alcohol use. The other type of psychotherapy we will use focuses on strengthening motivation to recover from cocaine and/or alcohol use, and on developing techniques to handle possible barriers to recovery. We seek to enroll 300 patients in the study.

ELIGIBILITY:
Inclusion Criteria::

* Male and females, 18-65 years old.
* Meets DSM-IV criteria for current diagnoses of cocaine and alcohol dependence, determined by the SCID.
* In the past 30 days, S used no less than $200-worth of cocaine and >15 standard alcohol drinks (avg)/week with at least 1 day of 4 or more drinks, determined by the TLFB--adapted to collect daily cocaine use.
* Successful completion of medical detoxification, i.e., 5 consecutive days of abstinence from cocaine and alcohol, via self-reports and negative urine toxicology screens.
* Lives a commutable distance to the TRC and agrees to follow-up visits.
* Understands and signs the consent.

Exclusion Criteria::

* Abstinent from cocaine or alcohol for 30 days prior to signing consent form. (S may have been institutionalized in the prior month and still be eligible if his/her cocaine and alcohol use that month met inclusion criteria.)
* Current DSM-IV diagnosis of any substance dependence other than cocaine, alcohol, nicotine, or cannabis determined by the SCID.
* Evidence of opiate use in the past 30 days, determined by self-report on the SCID or ASI, and/or by a urine drug screen that is positive for opiates at treatment entry.
* Current treatment with psychotropic medications (excluding short-term use of benzodiazepines for detoxification), including disulfiram.
* History of unstable or serious medical illness, including need for opioid analgesics.
* History of epilepsy or seizure disorder.
* Severe physical or medical illnesses such as AIDS, active hepatitis, significant hepatocellular injury as evidenced by elevated bilirubin levels, or elevated levels over 3.5x normal of aspartate aminotransferase (AST), and serum glutamic-pyruvic transaminase (SGPT).
* Current severe psychiatric symptoms, e.g., psychosis, suicidal or homicidal ideation or mania.
* Use of an investigational medication in the past 30 days.
* Female Ss who are pregnant, nursing, or not using a reliable method of contraception. [Note: Criteria 4-10 will be assessed via the medical exam plus results from lab tests.]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 1998-01; Primary Completion 2003-02 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Pettinati, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania- Treatment Research Center, Philadelphia, Pennsylvania, United States